CLINICAL TRIAL: NCT03298854
Title: The Diagnostic Performance of Skeletal 99mTc-MDP SPECT/CT in Patients With Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mohamed Fathy (Other)
Responsible Party: Sponsor-Investigator, Mohamed Fathy, Resident of Nuclear Medicine, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SPECT/CTinlowbackpain
Record Dates: First submitted 2017-09-23; First posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: 99mTc-MDP SPECT/CT — Delayed whole body images, using Symbia-T-Siemens dual headed gamma camera, will be obtained 2-3 hours after injection of 15-25 mCi of Tc-99m MDP (Methylene diphosphonate) followed by SPECT images of the lumbar spine and pelvis.

SUMMARY:
To evaluate the diagnostic performance (sensitivity, specificity, Negative and positive predictive value) of skeletal co-registered SPECT/CT imaging in the detection of the etiology of low back pain in adolescent and adult patients

DETAILED DESCRIPTION:
Low back pain(LBP) is extremely common. Though estimates vary widely, studies in developed countries report one year prevalence of 22-65% and lifetime prevalence up to 84%. (Walker, 2000) (1) The differential diagnosis for back pain is broad and includes degenerative disease, infection, inflammation, tumors and trauma(Zukotynski, Curtis et al. 2010) (2). The etiology of low back pain in young athletes differs from that seen in adults, with bony etiology being more common than disc-related disease(Matesan, Behnia et al. 2016) (3).

The American College of Physicians and the American Pain Society classify LBP into the following broad categories: nonspecific LBP, back pain potentially associated with radiculopathy or spinal stenosis, and back pain potentially associated with another specific spinal cause. Additionally, guidelines emphasize a focused history and physical examination, reassurance, initial pain management medications if necessary, and consideration of physical therapies without imaging in patients with nonspecific LBP. Duration of symptoms also helps guide treatment algorithms in patients with acute, sub-acute, or chronic LBP.(Chou, Qaseem et al. 2011) (4).

Many imaging modalities are available to the clinician and radiologist for evaluating LBP. Application of these modalities depends on the working diagnosis, the urgency of the clinical problem, and comorbidities of the patient. Radiographs of the lumbar spine are not routinely recommended in acute nonspecific LBP because they are of limited diagnostic value. Radiography is the initial imaging study of choice for assessing LBP in patients with a history of trauma and patients suspected of possible vertebral compression fracture.In addition, radiographs are recommended to evaluate a young patient for ankylosing spondylitis.(Jarvik, Gold et al. 2015) (5)

Patients with LBP lasting for >6 weeks having completed conservative management with persistent radiculopathic symptoms, may seek magnetic resonance imaging (MRI). Patients with severe or progressive neurologic deficit on presentation and red flags should be evaluated with MRI. Computed tomography (CT) scans provide superior bone detail but are not as useful in depicting soft tissue pathologies such as disc disease when compared with MRI. CT is useful for revealing bone structural problems such as spondylolysis, pseudarthrosis, fracture, scoliosis, and stenosis and for postsurgical evaluation of bone graft integrity, surgical fusion, and instrumentation (Brinjikji, Luetmer et al. 2015) (6)

Tc-99m methylene diphosphonates bone scan is a highly sensitive technique for detection of bone diseases and can allow the detection of the pathophysiology of trauma at a very early stage. Due its excellent sensitivity it is often used as a screening tool, however limited anatomical details result in poor specificity, It can be performed as limited or whole body bone scintigraphy (Van der Wall, Lee et al. 2010) (7). Dynamic and blood pool phases can increase specificity in the diagnosis of inflammatory pathology, but they are not routinely used in cases of facet joint disease (Shur, Corrigan et al. 2015) (8)

Bone scan is a useful clinical tool to explore the etiology of low back pain like spondylolysis and other less common etiologies in young athletes. It is also particularly important to detect the active source of pain when more than one bony abnormality is seen in anatomical imaging. The addition of three dimensional data acquisition SPECT (single photon emission computed tomography) increases the clinical accuracy due to increased contrast resolution and anatomical localization.(Matesan, Behnia et al. 2016) (3)

Radionuclide bone scintigraphy with (SPECT) provides functional imaging and is used to detect microcalcification due to increased osteoblastic activity. In the absence of other pathology the foci of increased osteoblastic activity reflect areas of mechanical stress and degenerative change in the skeleton. SPECT has been widely used to evaluate patients with spinal pain and facet joint arthropathy. For the detection of clinically significant facet arthropathy, The SPECT/CT images have an incremental diagnostic value that can influence clinical management by selecting only SPECT positive facet joint targets. (Matar, Navalkissoor et al. 2013) (9)

For some aspects, SPECT/ CT can be helpful even in a trauma setting. In particular, the combination of highly sensitive but nonspecific scintigraphy with non-sensitive but highly specific computed tomography makes it particularly useful in anatomically complex regions such as the pelvis and spine. From a trauma surgeon's point of view, the four main indications for nuclear medicine imaging are the detection of (occult) fractures, and the imaging of inflammatory bone and joint diseases, chronic diseases and postoperative complications such as instability of instrumentation or implants. which can consistently be found in a substantial number of patients (Scheyerer, Pietsch et al. 2014) (10), However its use as an appropriate imaging modality should be considered carefully given the increased radiation dose in young individuals with benign disease and low dose CT protocols should be used (Shur, Corrigan et al. 2015) (8)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients more than 18 years old
* Suffering from mechanical low back pain, either acute (less than 4 weeks), sub-acute (4 weeks up to 3 months) or chronic (more than 3 months)

Exclusion Criteria:

* Patients with known history of malignant disease
* Patients with previous history of lumbar spine surgery
* Patients with severe pain who cannot withstand the long duration of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
The Diagnostic Performance of Skeletal 99mTc-MDP SPECT/CT in Patients with Low Back Pain | 2years
  evaluate the diagnostic performance (sensitivity, specificity, Negative and positive predictive value) of skeletal co-registered SPECT/CT imaging in the assessment of low back pain in adolescent and adult patients

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AH Mekkawy, professor, Study Director — Assiut University